CLINICAL TRIAL: NCT07376317
Title: Optimization of Immunotherapy Treatment for Advanced Melanoma in the Context of the Public Brazilian Health System (OTIMAS)
Acronym: OTIMAS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Milena Mak, Milena Mak, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1957/2021
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Melanoma Metastatic; Melanoma Recurrent; Cutaneous Melanoma; Stage IV Melanoma
Keywords: Pembrolizumab; Optimization of immunotherapy treatment; advanced melanoma; cutaneous melanoma; metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200mg IV Q3W for one year (17 cycles)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patient will receive pembrolizumab 200mg IV Q3W for one year (17 cycles)

SUMMARY:
The OTIMAS study is a phase II trial designed to evaluate if the duration of one year of pembrolizumab immunotherapy for advanced metastatic melanoma has equivalent efficacy as the two-year duration of historical controls.

DETAILED DESCRIPTION:
The development of immune checkpoints inhibitors marked a new era in the treatment of melanoma patients. The use these therapies has more than doubled the expected median overall survival of patients with metastatic melanoma compared with chemotherapy At 5-year follow-up, the median overall survival of patients treated with nivolumab, an anti-PD-1 agent, was 37.3 months compared with 11.2 months in the group treated with dacarbazine, a chemotherapy agent, which represented a 50% reduction in the risk of death with a hazard ratio (HR) of 0.5 (95% CI, 0.40 to 0.63; P < .0001). However, these revolutionary therapies are accessible only to a minority of the Brazilian population, as chemotherapy remains the standard of care for patients with advanced melanoma treated by the Brazilian public health system (Sistema Único de Saúde - SUS), which covers more than 70% of the population.

No published study has specifically evaluated the optimal treatment time with immune checkpoint inhibitors. In studies with nivolumab, treatment was administered until progression or limiting toxicities, whereas in studies with another PD-1 inhibitor, pembrolizumab, treatment was administered for two years.

The OTIMAS study is a phase II trial designed to evaluate if the duration of one year of pembrolizumab immunotherapy for advanced metastatic melanoma has equivalent efficacy as the two-year duration of historical controls.

In this study, patients with advanced (metastatic or unresectable) cutaneous melanoma are treated with pembrolizumab 200mg every 3 weeks for a maximum duration of 12 months. Efficacy will be measured according to RECIST v1.1 criteria, with progression-free survival (PSF) in 24 months as the primary endpoint, compared to historical control. Additionally, the study will assess microRNAs as possible biomarkers in the responders. Other secondary analysis include: quality of life by EORTC QLC-C30 and EuroQol-3L and cost-effectiveness (12 versus 24 months) in the context of Brazilian health system.

This trial is being conducted at Institute of Cancer of the State of São Paulo (ICESP), with an estimated duration of four years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant melanoma (with confirmed histopathological diagnosis) stages III and IV not amenable to locoregional treatment or curative treatment
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2
* Up to 1 (one) line of prior treatment with palliative chemotherapy (monotherapy), with documented progression and no residual toxicities greater than grade 1 according to CTCAE
* Estimated life expectancy greater than 12 weeks
* Adequate renal function, defined as creatinine clearance estimated by the Cockcroft-Gault equation equal to or greater than 30 mL/min;
* Adequate liver function, defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels equal to or less than 2.0 times the upper limit of normal and total bilirubin less than 2 times the upper limit of normal;
* Hemoglobin greater than or equal to 8 g/dL; neutrophil count equal to or greater than 1,000/mm3; platelet count equal to or greater than 100,000/mm3;
* Ability to understand and adhere to study procedures;
* Age over 18 years;
* Absence of active treatment for the underlying disease, with the exception of the use of bisphosphonates;

Exclusion Criteria:

* Uncontrolled Central Nervous System (CNS) metastases: active symptomatic disease in the central nervous system, requiring doses of corticosteroids greater than the equivalent of 10 mg/day of prednisone. Patients previously submitted to local treatment, such as radiotherapy, will be eligible if they have demonstrated clinical stability in the 2 weeks prior to the start of treatment;
* Diagnosis of uveal or mucosal melanoma;
* Diagnosis of acral melanoma;
* Leptomeningeal disease
* Pregnancy; effective contraceptive methods should be recommended to women of childbearing age;
* Uncontrolled associated disease;
* Known active hepatitis B and C;
* HIV with detectable viral load or CD4<350;
* Active autoimmune disease with use of immunosuppressive therapy or history of autoimmune disease whose risk of recurrence is considered high by the investigator;
* More than one line of prior systemic therapy in the context of metastatic or advanced disease or prior use of polychemotherapy;
* Prior use of anti-PD-1 in the (neo)adjuvant setting;
* Concomitant active malignant neoplasia;
* History of malignant neoplasia in the last 5 years, with the exception of squamous cell carcinoma, basal cell carcinoma of the skin, in situ tumors, prostate adenocarcinoma gleason <=6;
* Infection with systemic involvement in the last 2 weeks;
* Use of corticosteroids in a dose equivalent to greater than 10 mg/d of prednisone on a continuous basis.
* History of solid organ transplantation under immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil